CLINICAL TRIAL: NCT03337243
Title: Effect of Implanting Allogenic Cytokines Derived From Human Amniotic Membrane (HAM) and Mesenchymal Stem Cells Derived From Human Umbilical Cord Wharton's Jelly (HUMCWJ) on Pain and Functioning of Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sport and Spine Rehab Clinical Research Foundation (Other)
Responsible Party: Principal Investigator, Gary Hieronimus, Doctor of Chiropractic, Scott Medical Health Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: StemCell
Record Dates: First submitted 2017-05-25; First posted 2017-11-08 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Knee Osteoarthritis; Knee Pain Chronic; Joint Disease; Arthritis; Osteo Arthritis Knee; Musculoskeletal Disease
Keywords: Stem Cell Injection; Cytokine; Wharton's Jelly; Stem Cells
MeSH Terms: conditions — Osteoarthritis, Knee; Joint Diseases; Arthritis; Musculoskeletal Diseases | interventions — ATF7IP protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HAM and HUMCWJ Injections (Group 1) (Experimental): Participants who self-select into the Group 1 (Immediate Treatment) will be scheduled to undergo the HAM and HUMCWJ injections to the OA affected knee at the same visit.
  Interventions: Procedure: HAM and HUMCWJ Injections
- Control (Group 2) (No Intervention): Participants who self-select into Group 2 will choose to delay their HAM and HUMCWJ injection to the OA affected knee for at least 3 months or choose not to have the injections at all. Participants will be asked to keep track of pain management and therapy throughout the 3 months.

INTERVENTIONS:
Procedure: HAM and HUMCWJ Injections — SURGENEX SurForce® (1cc) allograft placental based tissue matrix, will be injected using a 22 gauge, 2-inch needle. The injection site (medial, lateral, patellar) will be determined based on the side with the most joint space from the findings of the most recent x-rays. The Physician will insert the needle fully into the joint space and begin to expel the fluid. He will achieve a continuous injection flow as he withdraws the needle back out of joint space. Immediately following the SURGENEX SurForce® injection, an injection of Predictive Biotech CORECYTE(TM) (1 cc) allograft umbilical cord-derived Warton's Jelly tissue matrix will be administered. This will be done using the exact same protocol as the SURGENEX SurForce® injection.
  Arms: HAM and HUMCWJ Injections (Group 1)

SUMMARY:
The purpose of this study is to compare the pain, functioning and pain medication consumption of knee osteoarthritis (OA) patients who have allogenic cytokines derived from human amniotic membranes (HAM) and allogenic mesenchymal stem cells derived from human umbilical cord Wharton's Jelly (HUMCWJ) implanted into the affected knee with knee OA patients who self-select to be in a non-intervention control group.

DETAILED DESCRIPTION:
A total of 60 patients will be recruited from Scott Medical Health Center in Pittsburgh, PA. Inclusion criteria for the study are knee OA patients who are eligible for HAM and HUMCWJ therapy of their knee, no previous HAM or HUMCWJ therapy, between the ages of 50-85, independently residing in the community, no previously diagnosed cognitive decline or mental illness, and not taking pain medication more than once per week for a condition other than knee OA. Recruitment will be done in two parts as participants will self-select to participate in one of two study groups. All participants who elect to have the procedure done at the initial consultation, meet inclusion criteria, and agree to be in the study will be placed in Group 1. Participants who do not wish to have the procedure, meet inclusion and exclusion criteria, and agree to be in the study will be placed in Group 2. Those participants who are unsure about the procedure and need more time to decide will be contacted 2 weeks later and then group will be determined by their decision. All participants will be required to sign a written informed consent prior to data collection. Following written consent, all participants will undergo data collection (T0). At T0, participants will complete a demographic and medication use questionnaire, the Western Ontario and McMaster Universities Arthritis Index (WOMAC), knee survey, and be timed during a single trial of three functional tasks. Participants will also provide a pain rating while completing each of the functional tasks. Group 1 will then undergo HAMS injection to the OA affected knee immediately following the testing battery. Group 2 will delay the HAMS injection to the OA affected knee for at least 3 months or never receive the injection. All participants will complete T1 data collection approximately 4 weeks following completion of T0 data collection and T2 data collection approximately 3 months following completion of T0 data collection. The T1 and T2 data collections will use the same data collection procedures and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* knee OA patients who are eligible for HAM and HUMCWJ therapy of their knee, no previous HAM or HUMCWJ therapy, between the ages of 50-85, independently residing in the community, no previously diagnosed cognitive decline or mental illness, and not taking pain medication more than once per week for a condition other than knee OA

Exclusion Criteria:

* Allergy to or use of penicillin, streptomycin, emphotericin B or dimethylsulfoxide. DMSO allergies and any immunocompromised conditions will also be excluded

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
Change in Western Ontario and McMaster Universities Arthritis Index (WOMAC) over 3 months | Baseline (T0), 4 weeks (T1), 3 months (T2)
Change in pain during sit-to-stand over 3 months | Baseline (T0), 4 weeks (T1), 3 months (T2)
  Participants will perform as many sit-to-stand movements as they can in 30 seconds and then will rate pain
Change in pain during supine to upright over 3 months | Baseline (T0), 4 weeks (T1), 3 months (T2)
  Participants will perform a supine to upright movement as quickly as they can and then will rate pain
Change in pain during ascent/decent stairs over 3 months | Baseline (T0), 4 weeks (T1), 3 months (T2)
  Participants will ascend and decent 10 stairs as quickly as they can and then will rate pain

CONTACTS AND LOCATIONS:
Locations (1):
- Scott Medical Health Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No